CLINICAL TRIAL: NCT03137498
Title: Lidocaine Versus Ketorolac for the Management of Renal Colic
Brief Title: Lidocaine vs Ketorolac for Management of Renal Colic in the Emergency Department
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Brooklyn Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 902683
Record Dates: First submitted 2017-03-06; First posted 2017-05-02 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Renal Colic
Keywords: renal colic; lidocaine; ketorolac; acute pain
MeSH Terms: conditions — Renal Colic; Acute Pain | interventions — Lidocaine; Prilocaine; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind placebo-controlled randomized trial where blinding will be conducted and applied to the study investigator, physicians, and nursing staff providing care to the patient. An independent biostatistician will conduct a statistical analysis with blinded data. Only the pharmacists preparing the study interventions will be unblended to the study treatments. The pharmacists procuring the interventions will not be part of data collection or analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Experimental): Lidocaine 1.5mg/kg IVPB in 50ml normal saline over 10 minutes (active experimental) and normal saline 1ml intravenous push injection (placebo)
  Interventions: Drug: Lidocaine
- Ketorolac (Active Comparator): Ketorolac 30mg (1ml) intravenous push injection (active intervention) and Normal saline 50ml IVPB over 10 minutes (placebo)
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 1.5mg/kg IVPB in 50ml normal saline over 10 minutes x 1dose
  Other Names: Prilocaine
  Arms: Lidocaine
Drug: Ketorolac — Ketorolac 30mg (1ml) intravenous push injection x 1dose
  Other Names: Toradol
  Arms: Ketorolac

SUMMARY:
The hypothesis of the study is that lidocaine will be as effective as ketorolac in decreasing patient's perception of pain as measured by the 10 point Visual Analogue Scale (VAS). The aim of the study is to compare the safety & efficacy of lidocaine versus ketorolac for acute pain secondary to renal colic in the Emergency Department (ED).

DETAILED DESCRIPTION:
The hypothesis of the study is that lidocaine will be as effective as ketorolac in decreasing patient's perception of pain as measured by the 10 point Visual Analogue Scale (VAS). The aim of the study is to compare the safety & efficacy of lidocaine versus ketorolac for acute pain secondary to renal colic in the Emergency Department (ED). The primary endpoint is patient's perception of pain as described by the use of numeric rating scale (NRS) at 15 minutes after initial study interventions. The secondary endpoints are incidence of adverse events during the study period, patient perception of pain as described by the use of NRS at 0, 5, 15, 30, 45, 60, 75, 90 minutes after initial administration of study interventions, frequency and mean dose of rescue analgesic therapy needed at 0, 5, 15, 30, 45, 60, 75, 90 minutes, incidence of adverse events such as but would not be limited to: dizziness, perioral numbness, nausea, vomiting, arrhythmia [examples could be but are not limited to: atrial fibrillation, ventricular tachycardia, ventricular fibrillation), hypotension (≤90/60 mmHg), flushing, headache, tremors, ear pain, injection site reactions, disorientation, respiratory depression (respiratory rate less than 12bpm), oxygen saturation less than 90%)], the number of bedside ultrasounds for diagnosis conducted, the number of CT scans for diagnosis conducted, result of radiologic imaging (Ultrasound / Computerized Tomography), time to patient discharge from the initiation of study medication/placebo, patient satisfaction of pain control based on a Likert Scale, the number of patients who consumed an adjuvant pain medication for analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and older
* Presenting with acute generalized pain secondary to suspected or confirmed renal colic
* Describes pain to be greater than or equal to 3 out of 10 on the numeric rating scale (NRS)
* Provides informed consent.

Exclusion Criteria:

* Reported/documented allergy to lidocaine OR ketorolac (Toradol) OR morphine, corn, aspirin, ibuprofen
* Patients who are hemodynamically unstable as dictated by the medical resident or attending [(Heart rate not within 60-110bpm); (Respiratory rate not within 12-20 bpm); (Blood pressure not within 90/50 to 180/100); (Oxygen saturation not within 94-100%)]
* Patient with unwillingness to provide informed consent
* Patients with past medical history of cardiovascular disorders (examples include but are not limited to: myocardial infarction, ischemic heart disease, atrial fibrillation, heart blocks, Wolff-Parkinson-White syndrome, slow heart rate, bradycardia, coronary artery disease, QT prolongation)
* Past medical history of: liver dysfunction (ie: cirrhosis), chronic alcohol abuse, gastrointestinal bleed or recent gastrointestinal bleed (within past 5 days), renal dysfunction or disease, seizures (or currently actively receiving treatment for seizures), inflammatory bowel disease (or currently actively receiving treatment for inflammatory bowel disease), hepatitis (or currently actively receiving treatment for hepatitis).
* History of liver transplant
* Currently on dialysis
* Has acute heart, kidney, liver, respiratory failure or trauma
* In altered mental status
* In significant trauma, actively breastfeeding or pregnant
* Has language barriers who are unable to describe pain,
* Weighing at or over 130kg
* Has a blood pressure reading greater than 180/120 mmHg at triage,
* Previously enrolled to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2019-03-06 (Estimated); Study Completion 2019-03-06 (Estimated)

PRIMARY OUTCOMES:
Pain score at 15 minutes | at 15 minutes after initial study interventions
  Patient's perception of pain as described by the use of numeric rating scale (NRS) at 15 minutes after initial study interventions

SECONDARY OUTCOMES:
Adverse event-dizziness | throughout study period (90 minutes)
  incidence of dizziness throughout
Adverse event-perioral numbness | throughout study period (90 minutes)
  incidence of perioral numbness
Adverse event-nausea | throughout study period (90 minutes)
  incidence of nausea
Adverse event-vomiting | throughout study period (90 minutes)
  incidence of vomiting
Adverse event-arrhythmia | throughout study period (90 minutes)
  incidence of arrhythmia (atrial fibrillation, ventricular tachycardia, ventricular fibrillation)
Adverse event-hypotension | throughout study period (90 minutes)
  incidence of hypotension (≤90/60 mmHg)
Adverse event-flushing | throughout study period (90 minutes)
  incidence of flushing
Adverse event-headache | throughout study period (90 minutes)
  incidence of headache
Adverse event-tremors | throughout study period (90 minutes)
  incidence of tremors
Adverse event-ear pain | throughout study period (90 minutes)
  incidence of ear pain
Adverse event-injection site reactions | throughout study period (90 minutes)
  incidence of injection site reactions
Adverse event-disorientation | throughout study period (90 minutes)
  incidence of disorientation
Adverse event-respiratory depression | throughout study period (90 minutes)
  incidence of respiratory depression (respiratory rate less than 12bpm)
Adverse event-oxygen saturation less than 90% | throughout study period (90 minutes)
  incidence of oxygen saturation less than 90%
patient satisfaction of pain control based on a Likert Scale | throughout study period (90 minutes)
  based on a Likert Scale
the number of patients who consumed an adjuvant pain medication for analgesia. | throughout study period (90 minutes)
  the number of patients who consumed an adjuvant pain medication for analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie de Souza, MD, Study Chair — The Brooklyn Hospital Center
Locations (1):
- The Brooklyn Hospital Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No